CLINICAL TRIAL: NCT04075409
Title: An Open-Label, Parallel Group, Single-Center Study to Investigate the Pharmacokinetic, Safety, and Tolerability Profiles of Padsevonil in CYP2C19 Genotyped Healthy Male Japanese Study Participants
Brief Title: A Study to Test the Safety, and Tolerability of Padsevonil in Healthy Male Japanese Study Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UP0083; JapicCTI-194958 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Healthy Japanese Participants
Keywords: Padsevonil; CYP2C19; Healthy Japanese Participants; Pharmacokinetics
MeSH Terms: interventions — padsevonil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Extensive metabolizers (Experimental): Participants will receive assigned single and multiple doses of padsevonil.
  Interventions: Drug: Padsevonil
- Intermediate metabolizers (Experimental): Participants will receive assigned single and multiple doses of padsevonil.
  Interventions: Drug: Padsevonil
- Poor metabolizers (Experimental): Participants will receive assigned single and multiple doses of padsevonil.
  Interventions: Drug: Padsevonil

INTERVENTIONS:
Drug: Padsevonil — Padsevonil will be administered in predefined dosages.

SUMMARY:
The purpose of the study is to investigate the pharmacokinetics (PK) of padesevonil in CYP2C19 genotyped healthy male Japanese study participants.

ELIGIBILITY:
Inclusion Criteria:

* The study participant must be 20 to 55 years of age inclusive, at the time of signing the informed consent
* The study participant is overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* The study participant is of Japanese descent as evidenced by appearance and verbal confirmation of familial heritage
* The study participant has a body weight ≥50 kg and body mass index within the range [18 to 30] kg/m^2 (inclusive)
* The study participant is male

Exclusion Criteria:

* The study participant has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study, such as a history of schizophrenia, or other psychotic disorder, bipolar disorder, or severe unipolar depression. The presence of potential psychiatric exclusion criteria will be determined based on the psychiatric history collected at the Screening Visit
* The study participant has a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders, capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data
* The study participant has a history of unexplained syncope or a family history of sudden death due to long QT syndrome
* The study participant has a lifetime history of suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt), or has had suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the "Screening/Baseline" version of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening
* The study participant has alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) >1.0 x upper limit of normal (ULN)
* The study participant has bilirubin >1.0 x ULN (isolated bilirubin >1.0 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 %)
* The study participant has current or chronic history of liver disease or known hepatic or biliary abnormalities
* The study participant has any clinically relevant electrocardiogram (ECG) finding at the Screening Visit or at Baseline.
* The study participant has made a blood or plasma donation or has had a comparable blood loss (>450 mL) within the last 30 days prior to Screening. Blood donation during the study is not permitted

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 39 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Up0083 001, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, Individual Patient Data cannot be adequately anonymized and there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

REFERENCES:
- [Derived] Chanteux H, MacPherson M, Kramer H, Otoul C, Okagaki T, Rospo C, De Bruyn S, Watling M, Bani M, Sciberras D. Overview of preclinical and clinical studies investigating pharmacokinetics and drug-drug interactions of padsevonil. Expert Opin Drug Metab Toxicol. 2024 Aug;20(8):841-855. doi: 10.1080/17425255.2024.2373108. Epub 2024 Jul 9. PMID 38932723

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in September 2019 and concluded in December 2019.
Pre-assignment Details: Participant flow refers to the Safety Set.
Groups:
- Extensive Metabolizers: Extensive metabolizers (Participants confirmed with genotype *1/*1) received a single oral dose of padsevonil (PSL) 200 mg in the morning on Day 1 of the Single-dose Period. During the Multiple-dose Period, participants received PSL 100 mg twice a day (BID) on Day 6, PSL 200 mg BID from Day 7 to Day 9, PSL 200 mg in the morning on Day 10; PSL 100 mg in the evening on Day 10, and PSL 100 mg BID from Day 11 to Day 12 orally.
- Intermediate Metabolizers: Intermediate metabolizers (Participants confirmed with genotype *1/*2,*1/*3) received a single oral dose of PSL 200 mg in the morning on Day 1 of the Single-dose Period. During the Multiple-dose Period, participants received PSL 100 mg BID on Day 6, PSL 200 mg BID from Day 7 to Day 9, PSL 200 mg in the morning on Day 10; PSL 100 mg in the evening on Day 10, and PSL 100 mg BID from Day 11 to Day 12 orally.
- Poor Metabolizers: Poor metabolizers (Participants confirmed with genotype *2/*2, *2/*3, *3/*3) received a single oral dose of PSL 200 mg in the morning on Day 1 of the Single-dose Period. During the Multiple-dose Period, participants received PSL 100 mg BID on Day 6, PSL 200 mg BID from Day 7 to Day 9, PSL 200 mg in the morning on Day 10; PSL 100 mg in the evening on Day 10, and PSL 100 mg BID from Day 11 to Day 12 orally.
Period: Overall Study
Arm/Group | Extensive Metabolizers | Intermediate Metabolizers | Poor Metabolizers
Started | 13 | 13 | 13
Completed | 13 | 13 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS) which consisted of all enrolled participants who received at least 1 dose of Padsevonil (PSL).
Arm/Group | Extensive Metabolizers | Intermediate Metabolizers | Poor Metabolizers | Total Title
Number analyzed (Participants) | 13 | 13 | 13 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 13 | 39
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (6.6) | 32.5 (5.9) | 32.5 (7.7) | 30.9 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 13 | 13 | 13 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 13 | 13 | 13 | 39

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of a Single Dose Padsevonil
Description: Cmax is the maximum plasma drug concentration of PSL observed from pharmacokinetic samples taken at predefined time points.
Time Frame: Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours postdose (up to Day 3)
Population: The Pharmacokinetic Per-protocol Set (PK-PPS) was a subset of the Safety Set, consisting of those study participants who had no important protocol deviations affecting the PK parameters and for whom a sufficient number of samples were available to determine at least 1 PK parameter.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Poor Metabolizers (PK-PPS): Poor metabolizers (Participants confirmed with genotype *2/*2, *2/*3, *3/*3) received a single oral dose of PSL 200 mg in the morning on Day 1 of the Single-dose Period. During the Multiple-dose Period, participants received PSL 100 mg BID on Day 6, PSL 200 mg BID from Day 7 to Day 9, PSL 200 mg in the morning on Day 10; PSL 100 mg in the evening on Day 10, and PSL 100 mg BID from Day 11 to Day 12 orally. Participants formed the Pharmacokinetic Per Protocol Set (PK-PPS).
- Intermediate Metabolizers (PK-PPS): Intermediate metabolizers (Participants confirmed with genotype *1/*2,*1/*3) received a single oral dose of PSL 200 mg in the morning on Day 1 of the Single-dose Period. During the Multiple-dose Period, participants received PSL 100 mg BID on Day 6, PSL 200 mg BID from Day 7 to Day 9, PSL 200 mg in the morning on Day 10; PSL 100 mg in the evening on Day 10, and PSL 100 mg BID from Day 11 to Day 12 orally. Participants formed the Pharmacokinetic Per Protocol Set (PK-PPS).
- Extensive Metabolizers (PK-PPS): Extensive metabolizers (Participants confirmed with genotype *1/*1) received a single oral dose of PSL 200 mg in the morning on Day 1 of the Single-dose Period. During the Multiple-dose Period, participants received PSL 100 mg BID on Day 6, PSL 200 mg BID from Day 7 to Day 9, PSL 200 mg in the morning on Day 10; PSL 100 mg in the evening on Day 10, and PSL 100 mg BID from Day 11 to Day 12 orally. Participants formed the Pharmacokinetic Per Protocol Set (PK-PPS).
Arm/Group | Poor Metabolizers (PK-PPS) | Intermediate Metabolizers (PK-PPS) | Extensive Metabolizers (PK-PPS)
Number analyzed (Participants) | 13 | 13 | 13
ng/mL | 1029 [832.5 to 1272] | 833.6 [674.6 to 1030] | 721.3 [583.6 to 891.4]
Statistical Analysis 1: Comparison: Poor Metabolizers (PK-PPS) vs Extensive Metabolizers (PK-PPS); Point estimates for the geometric least squares (LS) means ratio and the respective 2-sided 90% Confidence Intervals (CIs) were computed using the LS means and the root mean squares of error, based on of the log-transformed data with subsequent exponential transformation; Test type: Other; ANOVA; The ANOVA model included genotype group as the fixed effects. The natural logs were taken of the dependent variables and were back-transformed; LS means ratio = 1.426, 90% CI 2-sided [1.112 to 1.830]
Statistical Analysis 2: Comparison: Poor Metabolizers (PK-PPS) vs Intermediate Metabolizers (PK-PPS); Point estimates for the geometric least squares (LS) means ratio and the respective 2-sided 90% CIs were computed using the LS means and the root mean squares of error, based on of the log-transformed data with subsequent exponential transformation; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; LS means ratio = 1.234, 90% CI 2-sided [0.9619 to 1.584]
Statistical Analysis 3: Comparison: Intermediate Metabolizers (PK-PPS) vs Extensive Metabolizers (PK-PPS); [analysis description as in outcome 1, analysis 2]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; LS means ratio = 1.156, 90% CI 2-sided [0.9008 to 1.483]

2. Primary Outcome: Area Under the Curve From 0 to t (AUC(0-t)) of a Single Dose Padsevonil
Description: AUC(0-t) is the area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration.
Time Frame: Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours postdose (up to Day 3)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Poor Metabolizers (PK-PPS) | Intermediate Metabolizers (PK-PPS) | Extensive Metabolizers (PK-PPS)
Number analyzed (Participants) | 13 | 13 | 13
h*ng/mL | 5988 [4976 to 7206] | 4645 [3860 to 5589] | 2823 [2346 to 3397]
Statistical Analysis 1: Comparison: Poor Metabolizers (PK-PPS) vs Extensive Metabolizers (PK-PPS); [analysis description as in outcome 1, analysis 2]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; LS means ratio = 2.122, 90% CI 2-sided [1.706 to 2.638]
Statistical Analysis 2: Comparison: Poor Metabolizers (PK-PPS) vs Intermediate Metabolizers (PK-PPS); [analysis description as in outcome 1, analysis 2]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; LS means ratio = 1.289, 90% CI 2-sided [1.037 to 1.603]
Statistical Analysis 3: Comparison: Intermediate Metabolizers (PK-PPS) vs Extensive Metabolizers (PK-PPS); [analysis description as in outcome 1, analysis 2]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; LS means ratio = 1.646, 90% CI 2-sided [1.323 to 2.046]

3. Primary Outcome: Area Under the Curve From Time 0 to Infinity (AUC) of a Single Dose Padsevonil
Description: AUC is the area under the plasma concentration-time curve from time zero to infinity.
Time Frame: Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours postdose (up to Day 3)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Poor Metabolizers (PK-PPS) | Intermediate Metabolizers (PK-PPS) | Extensive Metabolizers (PK-PPS)
Number analyzed (Participants) | 13 | 13 | 13
h*ng/mL | 6024 [5009 to 7245] | 4666 [3879 to 5611] | 2837 [2359 to 3412]
Statistical Analysis 1: Comparison: Poor Metabolizers (PK-PPS) vs Extensive Metabolizers (PK-PPS); [analysis description as in outcome 1, analysis 2]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; LS means ratio = 2.124, 90% CI 2-sided [1.709 to 2.639]
Statistical Analysis 2: Comparison: Poor Metabolizers (PK-PPS) vs Intermediate Metabolizers (PK-PPS); [analysis description as in outcome 1, analysis 2]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; LS means ratio = 1.291, 90% CI 2-sided [1.039 to 1.604]
Statistical Analysis 3: Comparison: Intermediate Metabolizers (PK-PPS) vs Extensive Metabolizers (PK-PPS); [analysis description as in outcome 1, analysis 2]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; LS means ratio = 1.645, 90% CI 2-sided [1.324 to 2.044]

4. Primary Outcome: Terminal Half-life (t1/2) of a Single Dose Padsevonil
Description: The t1/2 is the apparent terminal half-life. Geometric Means and Geometric Coefficient of Variations were only calculated if at least 2/3 of the parameters were properly determined parameters (i.e. non-calculated and non-flagged).
Time Frame: Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours postdose (up to Day 3)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Extensive Metabolizers (PK-PPS) | Intermediate Metabolizers (PK-PPS) | Poor Metabolizers (PK-PPS)
Number analyzed (Participants) | 13 | 13 | 13
hours | 5.018 (22.2) | 5.904 (21.3) | 6.138 (24.1)

5. Primary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of a Single Dose Padsevonil
Description: The tmax is the time to reach maximum plasma concentration.
Time Frame: Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours postdose (up to Day 3)
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Extensive Metabolizers (PK-PPS) | Intermediate Metabolizers (PK-PPS) | Poor Metabolizers (PK-PPS)
Number analyzed (Participants) | 13 | 13 | 13
hours | 2.000 [0.500 to 4.00] | 3.000 [1.00 to 6.00] | 3.000 [0.500 to 3.00]

6. Primary Outcome: Maximum Plasma Concentration (Cmax) of Padsevonil at Steady-state (ss)
Description: Cmax, ss is the maximum plasma concentration of PSL observed from pharmacokinetic samples, taken at predefined time point at a steady-state.
Time Frame: Day 10: Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after the morning dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Poor Metabolizers (PK-PPS) | Intermediate Metabolizers (PK-PPS) | Extensive Metabolizers (PK-PPS)
Number analyzed (Participants) | 13 | 13 | 13
ng/mL | 1375 [1154 to 1639] | 1318 [1106 to 1570] | 1263 [1060 to 1505]
Statistical Analysis 1: Comparison: Poor Metabolizers (PK-PPS) vs Extensive Metabolizers (PK-PPS); [analysis description as in outcome 1, analysis 2]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; LS means ratio = 1.089, 90% CI 2-sided [0.8859 to 1.339]
Statistical Analysis 2: Comparison: Poor Metabolizers (PK-PPS) vs Intermediate Metabolizers (PK-PPS); [analysis description as in outcome 1, analysis 2]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; LS means ratio = 1.044, 90% CI 2-sided [0.8489 to 1.283]
Statistical Analysis 3: Comparison: Intermediate Metabolizers (PK-PPS) vs Extensive Metabolizers (PK-PPS); [analysis description as in outcome 1, analysis 2]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; LS means ratio = 1.044, 90% CI 2-sided [0.8489 to 1.283]

7. Primary Outcome: Area Under the Curve Over a Dosing Interval (AUCtau) of Multiple Doses Padsevonil
Description: AUCtau is the area under the plasma concentration time curve over a dosing interval.
Time Frame: Day 10: Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after the morning dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Poor Metabolizers (PK-PPS) | Intermediate Metabolizers (PK-PPS) | Extensive Metabolizers (PK-PPS)
Number analyzed (Participants) | 13 | 13 | 13
h*ng/mL | 6482 [5435 to 7730] | 6488 [5441 to 7737] | 4824 [4045 to 5753]
Statistical Analysis 1: Comparison: Poor Metabolizers (PK-PPS) vs Extensive Metabolizers (PK-PPS); [analysis description as in outcome 1, analysis 2]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; LS means ratio = 1.344, 90% CI 2-sided [1.092 to 1.653]
Statistical Analysis 2: Comparison: Poor Metabolizers (PK-PPS) vs Intermediate Metabolizers (PK-PPS); [analysis description as in outcome 1, analysis 2]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; LS means ratio = 0.9991, 90% CI 2-sided [0.8120 to 1.229]
Statistical Analysis 3: Comparison: Intermediate Metabolizers (PK-PPS) vs Extensive Metabolizers (PK-PPS); [analysis description as in outcome 1, analysis 2]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; LS means ratio = 1.345, 90% CI 2-sided [1.093 to 1.655]

8. Primary Outcome: Terminal Half-life (t1/2) of Multiple Doses Padsevonil
Description: The t1/2 is the apparent terminal half-life.
Time Frame: Day 10: Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after the morning dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Extensive Metabolizers (PK-PPS) | Intermediate Metabolizers (PK-PPS) | Poor Metabolizers (PK-PPS)
Number analyzed (Participants) | 8 | 2 | 1
hours | NA (NA) — Half-life values could not be estimated for more than one third of the participants due to at least one of the reasons (data points < 3, Lambda_z interval < 2x half-life, or Adjusted R^2 < 0.8). | NA (NA) — Half-life values could not be estimated for more than one third of the participants due to at least one of the reasons (data points < 3, Lambda_z interval < 2x half-life, or Adjusted R^2 < 0.8). | NA (NA) — Half-life values could not be estimated for more than one third of the participants due to at least one of the reasons (data points < 3, Lambda_z interval < 2x half-life, or Adjusted R^2 < 0.8).

9. Primary Outcome: Time to Reach Maximum Concentration (Tmax) for Padsevonil at Steady-state (ss)
Description: The tmax, ss is the time of observed maximum plasma concentration at a steady-state.
Time Frame: Day 10: Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after the morning dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Extensive Metabolizers (PK-PPS) | Intermediate Metabolizers (PK-PPS) | Poor Metabolizers (PK-PPS)
Number analyzed (Participants) | 13 | 13 | 13
hours | 1.500 [0.500 to 4.00] | 2.000 [1.00 to 4.00] | 1.500 [0.500 to 3.00]

10. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events During the Study
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant or trial participant that is administered a drug or biologic (medicinal product) or that is using a medical device. The event does not necessarily have a causal relationship with that treatment or usage.
Time Frame: From Baseline until the Safety Follow-up Visit (up to Day 21)
Population: The Safety Set (SS) consisted of all study participants who had received at least 1 dose of padsevonil.
Measure: Number; unit: percentage of participants
Groups:
- Extensive Metabolizers Single Dose (SS): Extensive metabolizers (Participants confirmed with genotype *1/*1) received a single oral dose of PSL 200 mg in the morning on Day 1 of the Single-dose Period. Participants formed the Safety Set (SS).
- Intermediate Metabolizers Single Dose (SS): Intermediate metabolizers (Participants confirmed with genotype *1/*2,*1/*3) received a single oral dose of PSL 200 mg in the morning on Day 1 of the Single-dose Period. Participants formed the Safety Set (SS).
- Poor Metabolizers Single Dose (SS): Poor metabolizers (Participants confirmed with genotype *2/*2, *2/*3, *3/*3) received a single oral dose of PSL 200 mg in the morning on Day 1 of the Single-dose Period. Participants formed the Safety Set (SS).
- Extensive Metabolizers Multiple Dose (SS): Extensive metabolizers (Participants confirmed with genotype *1/*1) received PSL 100 mg BID on Day 6, PSL 200 mg BID from Day 7 to Day 9, PSL 200 mg in the morning on Day 10; PSL 100 mg in the evening on Day 10, and PSL 100 mg BID from Day 11 to Day 12 orally of Multiple-dose Period. Participants formed the Safety Set (SS).
- Intermediate Metabolizers Multiple Dose (SS): Intermediate metabolizers (Participants confirmed with genotype *1/*2,*1/*3) received PSL 100 mg BID on Day 6, PSL 200 mg BID from Day 7 to Day 9, PSL 200 mg in the morning on Day 10; PSL 100 mg in the evening on Day 10, and PSL 100 mg BID from Day 11 to Day 12 orally of Multiple-dose Period. Participants formed the Safety Set (SS).
- Poor Metabolizers Multiple Dose (SS): Poor metabolizers (Participants confirmed with genotype *2/*2, *2/*3, *3/*3) received PSL 100 mg BID on Day 6, PSL 200 mg BID from Day 7 to Day 9, PSL 200 mg in the morning on Day 10; PSL 100 mg in the evening on Day 10, and PSL 100 mg BID from Day 11 to Day 12 orally of Multiple-dose Period. Participants formed the Safety Set (SS).
Arm/Group | Extensive Metabolizers Single Dose (SS) | Intermediate Metabolizers Single Dose (SS) | Poor Metabolizers Single Dose (SS) | Extensive Metabolizers Multiple Dose (SS) | Intermediate Metabolizers Multiple Dose (SS) | Poor Metabolizers Multiple Dose (SS)
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13 | 13
percentage of participants | 100 | 100 | 100 | 100 | 100 | 100

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from Baseline until the Safety Follow-up Visit (up to Day 21)
Description: One participant could experience multiple adverse events.
Arm/Group | Extensive Metabolizers Single Dose (SS) | Intermediate Metabolizers Single Dose (SS) | Poor Metabolizers Single Dose (SS) | Extensive Metabolizers Multiple Dose (SS) | Intermediate Metabolizers Multiple Dose (SS) | Poor Metabolizers Multiple Dose (SS)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13 | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13 | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 13/13 | 13/13 | 13/13 | 13/13 | 13/13 | 13/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extensive Metabolizers Single Dose (SS) (N=13) | Intermediate Metabolizers Single Dose (SS) (N=13) | Poor Metabolizers Single Dose (SS) (N=13) | Extensive Metabolizers Multiple Dose (SS) (N=13) | Intermediate Metabolizers Multiple Dose (SS) (N=13) | Poor Metabolizers Multiple Dose (SS) (N=13)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 1 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 13 (13) | 13 (13) | 13 (14) | 13 (73) | 13 (78) | 13 (84)
Dizziness (Nervous system disorders) | 6 (6) | 9 (9) | 8 (9) | 7 (23) | 8 (28) | 8 (29)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 5 (7) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT04075409/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT04075409/SAP_001.pdf